CLINICAL TRIAL: NCT02739347
Title: Non-Invasive Direct Current Stimulation for Cognition in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit successfully
Sponsor: Baylor College of Medicine (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Raymond Cho, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-42322
Record Dates: First submitted 2016-04-05; First posted 2016-04-15 (Estimated); Results first posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-06

CONDITIONS: Schizophrenia; Psychosis
Keywords: tDCS; cognitive control; working memory; EEG; gamma oscillations
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Stimulation (Experimental): Active stimulation group will receive 20 min of 2 mA direct current stimulation.
  Interventions: Device: Active Trans-cranial direct-current stimulation
- Sham Stimulation (Sham Comparator): This will be an active sham involving brief (15 msec) low current (0.11 mA) pulses every 550 ms.
  Interventions: Device: Sham Trans-cranial direct current stimulation

INTERVENTIONS:
Device: Active Trans-cranial direct-current stimulation — Active stimulation group will receive 20 min of 2 mA direct current stimulation.
  Other Names: tDCS
  Arms: Active Stimulation
Device: Sham Trans-cranial direct current stimulation — This will be an active sham involving brief (15 msec) low current (0.11 mA) pulses every 550 ms.
  Other Names: tDCS
  Arms: Sham Stimulation

SUMMARY:
This study proposes to assess the effect of trans-cranial direct current stimulation (tDCS) on cognitive control, working memory, functional, clinical, and cognitive outcomes in schizophrenia patients.

DETAILED DESCRIPTION:
Cognitive functions and EEG correlates will be thoroughly assessed in schizophrenia patients undergoing a tDCS treatment and compared with patients receiving a placebo stimulation. The treatment will involve 20 minutes of tDCS application to the left prefrontal and temporo-parietal cortex, twice a day for five days, a procedure shown to be effective in improving other symptoms of psychosis such as negative symptoms and hallucinations. Critically, in addition to standard neuropsychological testing, cognitive assessments will involve tasks that tap cognitive control and working memory, impairments in which comprise two of the core cognitive disturbances in schizophrenia and which have been linked to brain rhythm disturbances measurable by EEG recordings. Investigators will also assess changes in functional outcome by tDCS and investigate relationships between improvements in cognition, brain rhythms and functional outcome. All these assessments will occur just prior to tDCS application, just after completion of the tDCS series, and then again at 2 months follow-up. There will be two separate independent groups of patients who will be randomized to active versus sham treatments. The first group will have early course schizophrenia (less than 5 years of antipsychotic treatment; n=40). The second group will be chronic schizophrenia (greater than 5 years of antipsychotic treatment; n=40).

Relevance

This proposal would be the first integrated study of the effects of tDCS on cognitive symptoms, brain function and functional outcome in schizophrenia. A positive outcome would represent a marked improvement in clinical therapeutics for cognition in psychosis and provide a powerful tool for improving functional outcome in this debilitating disorder. Understanding the impact on brain rhythm disturbances could support the study of similar stimulation-based therapeutic approaches to other neuropsychiatric disorders that shows similar disturbances in cognition and brain rhythms activity, such as bipolar disorder and autism.

ELIGIBILITY:
Inclusion Criteria:

Early course psychosis:

* DSM-V diagnosis of Schizophrenia, Schizoaffective disorder, or schizophreniform disorder.
* ages 18-50 years
* on stable doses of medication for at least one month
* not taking benzodiazepines or mood stabilizers.
* Mild to severe cognitive impairment in MATRICS Consensus Cognitive Battery (composite scores < 40)

Chronic psychosis:

Same as early course psychosis but >5 years of antipsychotic treatment

Exclusion Criteria:

* Diagnostic and Statistical Manual-Version V (DSM-V) diagnosis of mental retardation
* significant head injury
* medical illness affecting brain function or structure
* pregnancy or postpartum (<6 weeks after delivery or miscarriage)
* significant neurologic disorder (e.g seizure disorder)
* inability to provide informed consent
* significant color blindness that affects task performance
* Comorbidity for DSM-V substance abuse disorder within the past one month
* Temporal relation between illness onset and head injury
* Taking benzodiazepines or mood stabilizers (lithium allowed)
* Positive drug screen (excluding THC at baseline)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-05; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Cho, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be open to sharing after primary findings of study have been published.

REFERENCES:
- [Background] Brunelin J, Mondino M, Gassab L, Haesebaert F, Gaha L, Suaud-Chagny MF, Saoud M, Mechri A, Poulet E. Examining transcranial direct-current stimulation (tDCS) as a treatment for hallucinations in schizophrenia. Am J Psychiatry. 2012 Jul;169(7):719-24. doi: 10.1176/appi.ajp.2012.11071091. PMID 22581236
- [Background] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126
- [Background] Cho RY, Konecky RO, Carter CS. Impairments in frontal cortical gamma synchrony and cognitive control in schizophrenia. Proc Natl Acad Sci U S A. 2006 Dec 26;103(52):19878-83. doi: 10.1073/pnas.0609440103. Epub 2006 Dec 14. PMID 17170134
- [Background] Green MF. What are the functional consequences of neurocognitive deficits in schizophrenia? Am J Psychiatry. 1996 Mar;153(3):321-30. doi: 10.1176/ajp.153.3.321. PMID 8610818
- [Background] Lisman J, Buzsaki G. A neural coding scheme formed by the combined function of gamma and theta oscillations. Schizophr Bull. 2008 Sep;34(5):974-80. doi: 10.1093/schbul/sbn060. Epub 2008 Jun 16. PMID 18559405
- [Background] Mondino M, Brunelin J, Palm U, Brunoni AR, Poulet E, Fecteau S. Transcranial Direct Current Stimulation for the Treatment of Refractory Symptoms of Schizophrenia. Current Evidence and Future Directions. Curr Pharm Des. 2015;21(23):3373-83. doi: 10.2174/1381612821666150619093648. PMID 26088110
- [Background] Stagg CJ, Best JG, Stephenson MC, O'Shea J, Wylezinska M, Kincses ZT, Morris PG, Matthews PM, Johansen-Berg H. Polarity-sensitive modulation of cortical neurotransmitters by transcranial stimulation. J Neurosci. 2009 Apr 22;29(16):5202-6. doi: 10.1523/JNEUROSCI.4432-08.2009. PMID 19386916
- [Background] Stagg CJ, Nitsche MA. Physiological basis of transcranial direct current stimulation. Neuroscientist. 2011 Feb;17(1):37-53. doi: 10.1177/1073858410386614. PMID 21343407
- [Background] Uhlhaas PJ, Singer W. Abnormal neural oscillations and synchrony in schizophrenia. Nat Rev Neurosci. 2010 Feb;11(2):100-13. doi: 10.1038/nrn2774. PMID 20087360
- [Background] Volk DW, Lewis DA. Prefrontal cortical circuits in schizophrenia. Curr Top Behav Neurosci. 2010;4:485-508. doi: 10.1007/7854_2010_44. PMID 21312410

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The reason we have fewer subjects randomized than enrolled is that some participants did not meet criteria to be randomized. These subjects were consented and completed many assessments, but were ultimately not randomized due to how they scored on some assessments. For instance, some participants MCCB score was too high to be randomized into the study.
Pre-assignment Details: The primary reasons for ineligibility were not taking any anti-psychotic medication, and positive drug screen. There were also many who did not even enter screening due to the assessment that they would highly likely not meet the threshold of requirement cognitive impairment (MATRICS score < 40).
Period: Overall Study
Arm/Group | Active Stimulation | Sham Stimulation
Started | 5 | 7
Completed | 2 | 4
Not Completed | 3 | 3
Not completed — Adverse Event | 3 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10.2) | 33 (7.5) | 33 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Control
Description: The investigators will assess cognitive control using the Preparing to Overcome Prepotency (POP) task. The accuracy mean differences between the high and low control conditions will be used as dependent measures.
  The study is powered at 0.8 to observe a post-pre treatment improvement in cognitive control with a substantial effect size (d=0.56) compared to sham stimulation with effects relatively stable measured 2 months after baseline. The hypothesized effect size will be d=0.60.
Time Frame: Week 1
Population: We have reported all available data.
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Working Memory
Description: The investigators will assess working memory using a working memory task. The accuracy mean differences between the high and low control conditions will be used as dependent measures.
  The study is powered at 0.8 to observe a post-pre treatment improvement in cognitive control with a substantial effect size (d=0.56) compared to sham stimulation with effects relatively stable measured 2 months after baseline. The hypothesized effect size will be d=0.60.
Time Frame: Week 1
Population: We have reported all available data.
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Negative Symptoms
Description: A secondary outcome measure is the severity of negative symptoms as quantified by Scale for the Assessment of Negative Symptoms (SANS). This study is powered at 0.8 to observe a post-pre treatment improvement in negative symptoms with a moderate effect size (d=0.56) compared to sham stimulation with effects relatively stable measured 2 months after baseline. The hypothesized effect size will be d=0.60.
Time Frame: Week 1
Population: We have reported all available data.
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Auditory Hallucinations
Description: A secondary outcome measure is the change over time in the severity of auditory hallucinations as assessed by the Auditory Hallucination Rating Scale (AHRS).
  In a study conducted using a similar montage and current strength (Brunelin et. al 2012), a reduction in auditory hallucinations with a substantial effect size (d=1.58) was observed in 30 patients with schizophrenia. However, as their study recruited only those patients with severe hallucinations while the current study does not have such an inclusion criterion. The investigators expect a more modest effect size of d=0.60.
Time Frame: Week 1
Population: We have reported all available data.
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Two months.
Arm/Group | Active Stimulation | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 1/5 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation (N=5) | Sham Stimulation (N=7)
Minor Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Minor burn and itching at sight of tDCS electrodes
Cognitive Decline (Psychiatric disorders) | 0 (0) | 1 (1) — Cognitive decline related to schizophrenia

LIMITATIONS AND CAVEATS:
Despite concerted and exhaustive subject recruitment efforts, the total number of patients completing the protocol was minimal. As such the sample size was inadequate for deriving any meaningful descriptive statistics or statistical comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT02739347/Prot_SAP_000.pdf